CLINICAL TRIAL: NCT07016139
Title: The Relationship Between Core Stability, Extremity Proprioception, and Dynamic Balance in Young Adults
Brief Title: Core-Proprioception-Balance Link
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veysel Akduman, PhD., Harran University
Other Study IDs: 05.12.2016-106
Record Dates: First submitted 2025-05-16; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Core Stabilization; Proprioception; Dynamic Balance
Keywords: Core Endurance; Hip Joint; Postural Balance; Proprioception; Shoulder Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background/Objectives: Core muscular endurance is believed to support both postural control and proprioceptive accuracy. This study aimed to investigate the relationship between core endurance, dynamic balance, and proprioceptive function of the hip and shoulder joints in healthy young adults. Methods: Sixty healthy young adults (mean age: 20.9 ± 2.4 years) participated. Core endurance was evaluated using McGill tests: Trunk Anterior Flexor Test (TAFT), Trunk Posterior Extensor Test (TPET), Right and Left Lateral Plank Tests (RLPT, LLPT). Dynamic balance was assessed with the Pedalo® platform, while shoulder and hip proprioception (flexion and abduction) was measured using the Biodex System 3 Pro. Results: Significant positive correlations were observed among all McGill tests, especially between RLPT and LLPT (r = 0.803, p < 0.05). TPET showed significant negative correlations with shoulder proprioception (flexion and abduction, p < 0.05), indicating that higher core endurance may enhance proprioceptive acuity. TAFT and TPET were also positively associated with dynamic balance. Conclusions: These findings indicate that trunk flexor and extensor endurance contribute to dynamic balance, and TPET may also reflect proprioceptive capacity in the shoulder. Core endurance training may thus have value in both balance and sensorimotor rehabilitation.

DETAILED DESCRIPTION:
Introduction Core musculature comprises a complex anatomical structure, including the hips and pelvic floor at the base, the diaphragm superiorly, the oblique muscles laterally, the gluteal and paraspinal muscles posteriorly, and the abdominal muscles anteriorly. This integrated system plays a vital role in balancing biomechanical forces acting on the body, enhancing force production in the extremities, and optimizing movement efficiency. Furthermore, by surrounding the trunk, it contributes significantly to spinal stability and the maintenance of upright posture. The core muscles, which play a key role in stabilizing the trunk and pelvis, also constitute the center of the kinetic chain. Core muscles play a crucial role in transmitting energy and force from the proximal to the distal segments through this chain, facilitating effective force transfer to the extremities. These functions enhance peripheral joint stability and decrease the risk of injury during physical activity. Core stability is defined as the capacity to control trunk position and movement relative to the pelvis effectively, and it plays a pivotal role in maintaining postural control. The core is considered a functional unit comprising muscle groups that collaboratively contribute to spinal stabilization. This stability emerges through the integrated action of motor control systems and muscular strength. Enhanced core stability promotes efficient force transmission throughout the kinetic chain, increases trunk muscle endurance, and supports both static and dynamic balance performance.

Balance is defined as the ability to maintain a stable posture by regulating the body's position in space. While static balance refers to sustaining postural stability in the absence of external disturbances, dynamic balance involves the capacity to restore and preserve stability during or following voluntary movement. Both components of balance are closely associated with trunk stability and reflect the efficiency of postural control systems. Trunk stability refers to the capacity to maintain control of the trunk both at rest and during dynamic or fine motor tasks. This control relies on two fundamental yet interrelated mechanisms: maintaining the projection of the body's center of gravity within the base of support and aligning body segments along the vertical axis. Enhancing core muscle strength contributes to postural control by minimizing deviations in the center of mass and reducing trunk sway. The efficiency of this postural mechanism is strongly influenced by neuromuscular control.

Neuromuscular control is closely associated with the proprioceptive component of the sensorimotor system. Proprioception refers to the transmission of afferent signals from mechanoreceptors located in muscles, ligaments, facet joints, and intervertebral discs to the central nervous system. Among these structures, the paraspinal muscles, which contain a high density of muscle spindles, play a critical role in regulating trunk movements. Disruptions in the proprioceptive signaling pathway can impair the development of accurate motor patterns and reduce overall movement quality.

Despite extensive literature on core stability and postural control, the relationship between core endurance and proprioceptive acuity in the upper and lower extremities remains underexplored. Clarifying this association is of particular interest in both clinical rehabilitation and athletic performance contexts. Therefore, the present study aims to investigate the effects of core muscle endurance on proprioceptive function in the shoulder and hip joints, and to examine how these variables relate to dynamic balance performance in healthy young adults.

Materials and Methods Participants This study included 60 healthy volunteers (37 females, 23 males; mean age: 20.9 ± 2.46 years). In this study, the sample size was determined by considering both the findings from previous studies and the need to compensate for data losses and preserve statistical power. In a similar study in the literature, a regression analysis that investigated the association between core endurance and dynamic balance found R² = 0.24. Based on this value, when the effect size was estimated using the formula f² = R² / (1 - R²), f² = 0.31 was obtained. An a priori power analysis conducted using G*Power (α = 0.05, power = 0.80, 5 predictor variables) determined that a minimum of 48 participants was needed to detect this effect size. The sample was planned to consist of at least 60 people, considering a potential attrition rate of 25% during the data collection phase. After completing the study, researchers performed post hoc power analysis for core endurance tests and found the lowest R² value of 0.19 in regression analyses. Using this value, researchers calculated the effect size as 0.24 with the f² = R² / (1 - R²) formula researchers made. Given these data (α = 0.05, f² = 0.24; predictors = 5; n = 60), statistical power was confirmed to be 0.80. These results indicate that the sample size was sufficient both during the planning phase and upon post-hoc verification.

Inclusion criteria included volunteering to participate in the research and not having participated in any previous study involving core endurance, proprioception, or balance assessments. Exclusion criteria were the presence of any known neurological, orthopedic, cardiovascular, or pulmonary disorders; visual impairments that could affect postural or balance assessments; pregnancy; refusal to participate in the study; and reporting pain or discomfort during exercise.

Ethical approval was obtained from the Ethics and Research Committee of Marmara University, and the study was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all participants before inclusion. Assessments were conducted in the following sequence: core endurance, proprioception, and dynamic balance.

McGill Core Endurance Test Core endurance was assessed using the McGill test protocol, which includes four static positions: trunk anterior flexor, trunk posterior extensor, and left and right lateral planks. These tests have demonstrated high reliability.

The participants practiced once to find the correct position, and then the maximum time each participant could maintain the static position was recorded for each test. A single examiner conducted all tests, gave standardized start and stop commands, and determined the end of the test to ensure reliability. Test termination occurred if trunk alignment deviated more than 10° from the initial position. All timing was controlled using a stopwatch to maintain consistency. Tests were conducted in a randomized order, with 5-minute rest intervals between positions and 1-minute intervals between trials. The test order was randomized across participants.

Trunk Anterior Flexor Test (TAFT): Participants sat on a mat with knees bent at 90° and the trunk leaning back at 60°, both angles verified with a goniometer. Arms were crossed over the chest. The test ended when the trunk could no longer maintain the 60° angle.

Lateral Plank Tests (Left and Right): In the right lateral plank test (RLPT), participants supported themselves on the right elbow placed under the shoulder, with the left hand on the opposite shoulder. Feet were stacked. The test was terminated when trunk or lower extremity alignment was lost. The same procedure was followed for the left side (LLPT).

Trunk Posterior Extensor Test (TPET): In the prone position, participants' anterior superior iliac spines were aligned with the edge of a plinth. The upper body was unsupported, and hands initially rested on a chair before being crossed over the chest. The lower body was stabilized with straps above and below the knees. Timing began once hands were lifted and posture was held horizontally. The test ended when posture could no longer be sustained.

Dynamic Balance Dynamic balance was assessed using the Pedalo® balance platform, which evaluates postural control and balance by monitoring center of pressure oscillations. Participants stood on the platform and attempted to maintain balance for one minute. Oscillations were recorded for analysis.

Proprioception Flexion and abduction movements of the shoulder and hip were selected for proprioception assessment due to their established reliability and clinical relevance. Proprioceptive errors during these movements are consistently linked to general joint position sense and functional deficits, making them valuable indicators of global proprioceptive function. The consistency and reliability of flexion and abduction measurements, combined with their clinical relevance, suggest these measurements are sufficient for assessing proprioception in both the shoulder and hip joints. The Biodex System 3 Pro Multi-Joint System® (Biodex Medical Inc., Shirley, NY, USA) was used to assess proprioception, offering high reliability across multiple joints. According to the manufacturer, there is no significant difference in proprioceptive assessment between Biodex Systems III and IV.

Active joint position sense (JPS) of the dominant shoulder and hip was assessed in flexion and abduction. The range of motion (ROM) for each movement was initially measured using a standard goniometer. Target angles were then set at 50% of the individual ROM, as proprioceptive errors are typically more pronounced at lower joint angles. Anthropometric adjustments (e.g., seat height, lever arm length) were made according to the operational guidelines of the Biodex system. Participants were first familiarized with the target angle via three open-eye trials. Then, with eyes closed, each participant actively reproduced each angle three times. The mean of the trials was used for analysis.

Statistical Analysis All statistical analyses were performed using IBM SPSS Statistics version 22.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics were expressed as mean ± standard deviation (SD), along with minimum and maximum values. Normality of data was evaluated using the Shapiro-Wilk test. Pearson correlation analysis was used to determine the relationships between core endurance scores (Trunk Flexor, Lateral Plank Left & Right, Trunk Extensor), dynamic balance, and joint proprioception (hip and shoulder abduction and flexion). A p-value < 0.05 was considered statistically significant. Correlation coefficients (r) were interpreted as follows: weak (0.10-0.39), moderate (0.40-0.69), and strong (0.70-1.00).

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study
* Provided written informed consent
* No prior participation in studies involving:

  * Core endurance assessment
  * Proprioception assessment
  * Balance assessment

Exclusion Criteria:

* Known neurological disorders
* Known orthopedic disorders
* Known cardiovascular disorders
* Known pulmonary disorders
* Visual impairments that may affect posture or balance
* Pregnancy
* Refusal to participate
* Reporting pain or discomfort during exercise

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study included 60 healthy volunteers (37 females, 23 males; mean age: 20.9 ± 2.46 years).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Regression Model Predictors for Core Endurance Tests to Proprioception and Balance | Immediately following recruitment
  This outcome measure evaluates the association between performance in core endurance tests (TAFT, TPET, RLPT, and LLPT) and proprioceptive and balance parameters, including shoulder flexion, shoulder abduction, hip flexion, and hip abduction angles. Multiple linear regression models will be used to assess the predictive value of each core test. Outcome metrics will be recorded in degrees (for joint angles) and balance scores from the Pedalo® platform.

SECONDARY OUTCOMES:
Correlation between McGill's core endurance tests | Immediately after all endurance tests are completed
  This outcome measure evaluates the relationship among performance scores from four McGill Core Endurance Tests: Trunk Anterior Flexor Test (TAFT), Trunk Posterior Extensor Test (TPET), Right Lateral Plank Test (RLPT), and Left Lateral Plank Test (LLPT). Statistical analysis will include bivariate correlation testing to assess potential linear relationships between endurance durations across the four test positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and lack of participant consent for data sharing beyond the scope of the original study.